CLINICAL TRIAL: NCT05930340
Title: Clinical Characteristics, Outcomes and Risk Factors for Mortality in Pregnant/Puerperal Women With COVID-19 Admitted to ICU in Turkey: a Multicenter, Retrospective Study From a Middle-income Country.
Status: Completed | Type: Observational
Sponsor: Turkish Intensive Care Society (Other)
Responsible Party: Principal Investigator, Nur Baykara, Prof.Dr., Kocaeli University
Other Study IDs: KÜ GOKAEK-2021/23.27
Record Dates: First submitted 2023-06-26; First posted 2023-07-05 (Actual); Last update posted 2023-07-05 (Actual); Status verified 2023-07

CONDITIONS: Key Words:COVID-19; Pregnancy; Intensive Care Unit; SARS-CoV-2; Mortality

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
We performed a national, multicenter, retrospective, cohort study. The study was announced on the Turkish Society of Intensive Care Medicine website, which included the study protocol, and the directors of ICUs caring for COVID-19 patients were invited. The study population comprised all SARS-CoV-2-infected pregnant or puerperal women (up to 6 weeks after birth) who were admitted to participating ICUs between 1 March 2020 and 1 January 2022. The exclusion criteria were patients aged <18 years old, patients with negative COVID-19 PCR test results, patients with active malignant disease, and organ transplant recipients.The following data were collected: patient demographics, gestational age or postpartum day on admission, date of ICU admission, comorbidities, vaccination status, Acute Physiology and Chronic Health Evaluation II (APACHE-2) and Sequential Organ Failure Assessment (SOFA) scores on admission, the worst SOFA score during the ICU stay, the ratio of lung infiltrates if diagnostic imaging was performed, the time interval from the start of symptoms to ICU admission, the duration of ICU stay, laboratory values on admission and the worst laboratory values during the ICU stay, the development of extrapulmonary organ injury,the presence of non-COVID-19 infections, The worst PaO2/FiO2 ratio during the ICU stay, the most invasive respiratory support method applied, and therapies were also recorded. Immunomodulatory therapies such as corticosteroids, IL inhibitors, intravenous immunoglobulin (IVIG) and cytokine hemadsorption, were also recorded. Fetal and neonatal complications were collected. LASSO regression and multiple logistic regression analyses were used to identify risk factors for maternal ICU mortality.

ELIGIBILITY:
Inclusion Criteria:

* The study population comprised all SARS-CoV-2-infected pregnant or puerperal women (up to 6 weeks after birth) who were admitted to participating ICUs between 1 March 2020 and 1 January 2022.

Exclusion Criteria:

* Patients aged <18 years old, patients with negative COVID-19 PCR test results, patients with active malignant disease, and organ transplant recipients.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All SARS-CoV-2-infected pregnant or puerperal women (up to 6 weeks after birth) who were admitted to participating ICUs between 1 March 2020 and 1 January 2022.
Sampling Method: Probability Sample
Enrollment: 597 (Actual)
Dates: Start 2022-03-15 (Actual); Primary Completion 2022-07-30 (Actual); Study Completion 2022-07-30 (Actual)

PRIMARY OUTCOMES:
Maternal Mortality in ICU | Prognosis of pregnant/puerperal women with COVID-19 admitted to ICU

CONTACTS AND LOCATIONS:
Locations (1):
- Kocaeli University, Kocaeli, Turkey (Türkiye)